CLINICAL TRIAL: NCT03393507
Title: A Study of Apatinib in Combination With Chemotherapy Versus Chemotherapy Alone for Advanced Ovarian Cancer
Brief Title: A Study of Apatinib Treatment in for Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The People's Hospital of Leshan (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhang Xuan, M.D., head of the department of the obstetrics and gynecology, The People's Hospital of Leshan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS-OV-2018
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer; Chemotherapeutic Toxicity
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib combine with chemotherapy (Experimental)
  Interventions: Drug: Apatinib; Drug: Taxus + platinum
- chemotherapy (Active Comparator)
  Interventions: Drug: Taxus + platinum

INTERVENTIONS:
Drug: Apatinib — 500mg,po, adjusted to 250mg if cannot tolerate, 3 weeks a cycle for a total of 6 cycles
  Arms: apatinib combine with chemotherapy
Drug: Taxus + platinum — Taxanes are paclitaxel or docetaxel, and platinum is carboplatin or cisplatin. Docetaxel injection dose size of 60-75mg / m2, infusion time of 1 hour; paclitaxel injection dose size 135-175mg / m2, infusion time> 3 hours; injection of carboplatin dose according to the standard formula Calculated, AUC = 4-5, continued intravenous infusion the next day; cisplatin injection dose size of 75-100mg / m2.

SUMMARY:
The study is evaluated the effacy and safety of apatinib combined with chemotherapy in the advanced ovarian cancer

DETAILED DESCRIPTION:
Ovarian cancer and fallopian tube cancer are common gynecological malignancies in our country. Ovarian cancer ranks the second in the incidence of gynecologic malignancies. The mortality rate is the highest. The following three major characteristics exist: First, 70% of the patients are advanced patients; 70% of the patients Easy to relapse after treatment; Third, 5-year survival rate of about 30%, a serious threat to women's health. Our hospital ovarian cancer, tubal cancer patients because of regional constraints, the economy is poor, the more the past, the use of simple chemotherapy, relapse rate and mortality were higher.

In the latest National Comprehensive Cancer Network (NCCN) guidelines, bevacizumab plus CP is recommended for patients with stage II, III, and IV ovarian cancer and fallopian tube cancer, and clinical trials of new drugs are recommended for recurrent / metastatic ovarian cancer. Apatinib mesylate is a small molecule VEGFR tyrosine kinase inhibitor authored by Jiangsu Hengrui Pharmaceutical Co., Ltd., whose chemical name is N- [4- (Cyanocyclopentyl) phenylmethane sulfonate ] [2 - [(4-picolyl) amino] (3-pyridyl)] carboxamide of the formula C25H27N5O3S with a molecular weight of 493.58 (mesylate salt).Apatinib can effectively inhibit VEGFR-2 at a very low concentration, while higher concentrations can inhibit the action of apatinib, such as platelet-derived growth factor receptor (PDGFR), c-Kit and c- The site is the intracellular ATP binding site of the protein tyrosine receptor. Pharmacodynamic studies show that apatinib can inhibit the VEGFR-2 tyrosine kinase activity, blocking VEGF signaling after binding, resulting in inhibition of tumor angiogenesis. Preclinical studies have shown that apatinib has a strong inhibitory effect on the growth of many human nude mice xenografts such as sarcoma, colorectal cancer, non-small cell lung cancer, gastric cancer and liver cancer and is a broad-spectrum anti-tumor drug.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as epithelial ovarian cancer, fallopian tube cancer, stage II-IV period, the expected survival of> 6 months;
* ECOG <2;
* Liver and kidney function is normal;
* No uncontrollable high blood pressure, bleeding, perforation, obstruction.

Exclusion Criteria:

* Serious cardiopulmonary insufficiency, can not tolerate chemotherapy;
* Pregnant or lactating women;
* 3 years have occurred in other tumors (cervical cancer in situ, has cured basal cell carcinoma, except for bladder epithelial tumors);
* Allergic to apatinib or its accessories.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female can be enrolled
Enrollment: 34 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS(Progress free survival) | 24 month
  he length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
carcinoma antigen 125 (CA125) | 24month
  Cancer antigen 125 (CA-125) is a protein found on the surface of many ovarian cancer cells. It also can be found in other cancers and in small amounts in normal tissue. A CA-125 test measures the amount of this protein in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang xuan, Leshan, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided